CLINICAL TRIAL: NCT02438956
Title: Oral Glutathione Supplementation in Older Healthy Adults and Its Effect on the Number of Healthy Days Experienced During Four Months of Supplementation Compared to Placebo
Acronym: GSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Kyowa Hakko Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201500236
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Improvement in Immune Cell Function in Elderly Humans

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalline Cellulose (Placebo Comparator): looks like and is given in the same way as the experimental treatment but contains no active ingredient
  Interventions: Dietary Supplement: Crystalline Cellulose
- Glutathione supplement (Experimental): 500 mg/day Setria glutathione supplement
  Interventions: Dietary Supplement: Setria glutathione supplement

INTERVENTIONS:
Dietary Supplement: Setria glutathione supplement — 500 mg/day capsule taken in the morning for 120 days.
  Other Names: Setria
  Arms: Glutathione supplement
Dietary Supplement: Crystalline Cellulose — 500 mg/day capsule taken in the morning for 120 days.
  Other Names: Placebo
  Arms: Crystalline Cellulose

SUMMARY:
A randomized, double blind placebo-controlled parallel intervention in adults over the age of 50 will be performed. Participants will receive a supplement capsule containing placebo (Crystalline Cellulose) or 500mg of Setria® Glutathione to eat for 120 days. Glutathione is hypothesized to replenish the body's reserves that may be depleted through natural aging process, poor diet, or due to the detoxification process for drugs. The primary end point is the number of healthy days experienced during the duration of the study. Secondary endpoints include cellular and biochemical measures from blood samples taken before and after the study.

DETAILED DESCRIPTION:
The long term goal of this investigation is to understand how food components improve immune function, both in its ability to respond to pathogens and its ability to turn off when the response is no longer needed. The goal of this application is to examine mechanisms by which glutathione improves immune cells after consumption. The central hypothesis is that glutathione improves redox status within the cell, thereby improving cell function and increasing the number of healthy days experienced by the participants.

After obtaining informed consent, human participants will receive 500 mg/day of Setria® Glutathione or placebo for 120 days. Peripheral blood mononuclear cells (PBMC), neutrophils and serum will be obtained from blood draws before and after the 120 days. A daily diary of illness will be kept by each participant and will record any incidence of illness, the number of symptoms per incidence, and the number of days in which symptoms are present. This study is powered on the basis that over 120 days, the glutathione-supplemented group would experience 3% more healthy days compared to the placebo group. The analysis indicated 60 people per group.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* must have had at least one cold during the previous year
* age 50-75
* must discontinue other dietary supplement use

Exclusion Criteria:

* on arthritis medication
* on hypertension medication
* severe allergies
* compromised immune system
* high cholesterol, heart failure, angina, etc.
* diagnoses of diabetes or metabolic syndrome

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Severity and frequency of Cold / Flu symptoms | 120 days
  Participants will record any cold / flu symptoms in log throughout the study duration

SECONDARY OUTCOMES:
Improvement of immune cell function | 120 days
  Increased neutrophil respiratory burst; IFN-gamma and other cytokine production measurements; gd-T cell proliferation in mitogen-stimulated ex vivo culture

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Percival, PhD, Principal Investigator — University of Florida
Locations (1):
- 449 Food Science and Human Nutrition Department, University of Florida, Gainesville, Florida, United States